CLINICAL TRIAL: NCT00216411
Title: A Prospective Phase IV, Multicentre, Placebo-controlled Study to Demonstrate Changes in the Quality of Life Following DYSPORT Intramuscular Injection in the Treatment of Upper Limb Spasticity in Adult Post-Stroke Patients
Brief Title: Effects on Quality of Life Following Dysport Treatment in Post-stroke Spasticity of the Arm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-9B-52120-097
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Cerebrovascular Accident; Muscle Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dysport (Experimental)
  Interventions: Biological: Botulinum toxin type A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Dysport
Drug: Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the effect on Quality of Life of two cycles of Dysport treatment on post-stroke spasticity of the upper limb. The effect of treatment on spasticity and function will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* The patient has suffered a stroke, as defined by the World Health Organisation (WHO) criteria, at least 6 months previously.
* The patient has a hemiparetic arm and meets minimum score requirements on the Modified Ashworth Scale.
* The patient has the cognitive and communication ability to participate in the study.

Exclusion Criteria:

* Patients who have received botulinum toxin treatment within the past 120 days.
* Contraindication to botulinum toxin treatment.
* Patients who are receiving oral anti-spasticity medication and who have had a change in dosage of this medication in the month prior to study entry.
* Patients who have previously been treated with phenol for their upper limb spasticity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2004-11; Primary Completion 2006-07-20 (Actual); Study Completion 2006-07-20 (Actual)

PRIMARY OUTCOMES:
Change in quality of life measured using the Assessment of Quality of Life questionnaire (12 question version).

SECONDARY OUTCOMES:
Change in muscle spasticity assessed on Modified Ashworth Scale (MAS)
Change in the Modified Motor Assessment Scale
Change in patient disability and carer burden rating scale total score
Achievement of the patient identified functional outcome measures (Goal Attainment Scaling)
Change in the degree of pain
Change in depression rating scale total score
Global assessment of benefit

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (6):
- Australia (6):
  - St Josephs Hospital, Auburn, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Caulfield General Medical Centre, Caulfield, Victoria
  - Austin Health, Heidelberg, Victoria

REFERENCES:
- [Derived] Turner-Stokes L, Baguley IJ, De Graaff S, Katrak P, Davies L, McCrory P, Hughes A. Goal attainment scaling in the evaluation of treatment of upper limb spasticity with botulinum toxin: a secondary analysis from a double-blind placebo-controlled randomized clinical trial. J Rehabil Med. 2010 Jan;42(1):81-9. doi: 10.2340/16501977-0474. PMID 20111849